CLINICAL TRIAL: NCT03550703
Title: Open Label Phase II Clinical Trial of Myoma Immunotherapy
Brief Title: Open Label Immunotherapy of Myoma
Acronym: V3-myoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myoma01
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-05

CONDITIONS: Myoma;Uterus; Fibroid Uterus; Leiomyoma; Fibroma
MeSH Terms: conditions — Myofibroma; Leiomyoma; Fibroma

STUDY DESIGN:
Intervention Model Description: open label, single arm study
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm receiving V3-Myoma (Experimental): A single oral pill of V3-Myoma therapeutic vaccine containing pooled antigens circulating in peripheral blood and within myoma tissues
  Interventions: Biological: V3-Myoma

INTERVENTIONS:
Biological: V3-Myoma — Once daily oral pill of V3-Myoma

SUMMARY:
Myoma of the uterus or uterine fibroids are benign tumors that appears in the myometrium or the muscular layer of the uterus. It is one of the most common diseases in pre-climax women, reaching 12-25% of all gynecological diseases. There is an opinion that the true prevalence of myoma is much larger and reaches up to 80%, i.e., practically every second woman has it, often without knowing about. For the treatment of MM, surgical removal of the nodes or removal of the uterus is used. In addition, GnRH-agonist therapy is practiced, as well as embolization to block blood flow in the tumor. We propose to evaluate the immunotherapy approach in an open label Phase II study in 20 women with myoma, for whom no alternative therapy is available.

DETAILED DESCRIPTION:
Myoma or uterine fibroids are one of the most common gynecological diseases, which occurs in at least one third of women older than 35 years, and after 40 - in every second. We will test a new tablet preparation, V3-Myoma, obtained from hydrolyzed, inactivated blood and tumor tissues of patients with uterine myoma. When administered orally, V3-Myoma should cause a specific anti-tumor immune response and an anti-inflammatory effect. Such an effect is due to the phenomenon known in immunology, called oral tolerance, leading to a reduction in tumor mass and a decrease in inflammation. An important advantage of our approach is the absence of any negative side effects. In the next three month, we will conduct Phase II open label clinical study of this intervention in 30 women with confirmed diagnosis of myoma.

ELIGIBILITY:
Inclusion Criteria:

diagnosed myoma with single or multiple tumors presence of typical clinical symptoms associated with myoma -

Exclusion Criteria:

other gynecological diseases not related to myoma hysterectomy

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Myoma is a female health problem
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in tumor size compared to baseline | Once monthly for three months
  This parameter will be evaluated by pelvic examination and transvaginal ultrasonography

SECONDARY OUTCOMES:
Changes in bleeding pattern at and between menstruations | During and between periods for three months
  Self-evaluated by patient
Changes in level of pain associated with myoma, low back and legs, pelvic pressure and pain, if any | 3 months
  Self evaluated by patient
Changes in frequent urination or difficulty in emptying the bladder or constipation | 3 months
  Self evaluated by patient

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbaiar, PhD, MD/PhD, Study Chair — Immunitor LLC
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No
Upon study completion the data will be available in peer-reviewed publication